CLINICAL TRIAL: NCT01484834
Title: Comparison of Interventions to Promote Health in Workers: A Cluster Randomized Controled Trial
Brief Title: Comparison of Interventions to Promote Health in Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Antonio Jose Grande, Principal Investigator, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UMetodistaPiracicaba-2011
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-05

CONDITIONS: Health Behavior
Keywords: Physical Activity; Occupational Health; Quality of Life; Health Promotion
MeSH Terms: conditions — Health Behavior; Motor Activity | interventions — Exercise; Educational Status; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Exercise and Education (Experimental): Company A received intervention of exercise in the workplace, posters with tips on health and quality of life computer software. The interventions with physical exercise in the workplace, were performed in the morning shift and had duration of three months with 15 minutes each and were applied three times per week every other day. In order to keep the workers motivated and participating in the exercise in the workplace, the sessions were very varied, using broomstick, latex tubes, exercises in pairs, massage, sitting exercises and relaxation on mats.
  Interventions: Behavioral: Exercise and Education
- Exercise (Active Comparator): The intervention with physical exercise in the workplace, were performed in the morning shift and had duration of three months with 15 minutes each and were applied three times per week every other day. In order to keep the workers motivated and participating in the exercise in the workplace, the sessions were very varied, using broomstick, latex tubes, exercises in pairs, massage, sitting exercises and relaxation on mats.
  Interventions: Behavioral: Exercise
- Educational Intervention (Active Comparator): This company received a quality of life software and poster intervention with tips on health lifestyle. The posters were printed in A3 paper and eight of them were put up per month in different parts of the companies (near water fountains, rest places, cafeterias, near the restrooms and change rooms). The used messages, both by the posters and the software were basedon scientific evidence related to quality of life and health
  Interventions: Behavioral: Educational Intervention
- Control Company (Placebo Comparator): No intervention
  Interventions: Other: Control Company

INTERVENTIONS:
Behavioral: Exercise and Education — Exercise were prescribed three times a week with duration of fifteen minutes for three months.
  Educational Intervention were composed by a quality of life computer software and poster with tips on health behaviors
  Other Names: Worksite interventions; Physical activity at the workplace
  Arms: Exercise and Education
Behavioral: Exercise — Exercise were prescribed three times a week with duration of fifteen minutes for three months.
  Other Names: Worksite interventions; Physical activity at the workplace
  Arms: Exercise
Behavioral: Educational Intervention — This company received a quality of life software and poster intervention with tips on health lifestyle. The posters were printed in A3 paper and eight of them were put up per month in different parts of the companies (near water fountains, rest places, cafeterias, near the restrooms and change rooms). The used messages, both by the posters and the software were basedon scientific evidence related to quality of life and health
  Other Names: Worksite interventions; Physical activity at the workplace
  Arms: Educational Intervention
Other: Control Company — No intervention was applied for the participants of this group
  Arms: Control Company

SUMMARY:
The goal of this research was to investigate different intervention strategies in the workplace and their impact on quality of life of workers from companies in the city of Londrina, Parana, Brazil.

The interventions were composed by exercise in the workplace and educational interventions.

DETAILED DESCRIPTION:
The workplace has special features about human behaviors. Studies (Shepard 1996, Pratt 2008) has shown that workers participate of this kind of health promotion programs for various reasons: One reason is the convenience of doing something without having to look for it; another reason is group support, many workers who share difficulties due to their working demands can find support in each other, so that they could change health behavior. Furthermore there are patterns of formal and informal communication that can contribute to help more people to become healthier making their environment better. Finally, the norms of a corporate behavior can unite the group of workers seeking same objectives.

Additionally the literature has shown that adults increased workload, job insecurity and pressure to perform tasks (Sparks 1997). These facts has been shown that workplace is different from community based interventions and leisure interventions.

The outcomes proposed to study are different from other studies since the interventions focus changes in behaviors. Sedentary behavior has shown to have 23% of deaths from major chronic disease (WHO 2002).

As the populations rises around the world and with the prolonged life expectancies, the number of people with chronic diseases will raise (WHO 2006). By having positive changes in health behavior the costs of public health can be reduced. Studying different types of interventions and testing its efficacy in different places can help the policy makers to create healthier environments.

There are strategies being developed in the workplace, but its efficacy is being challenged. There are some researches that show no evidence to prove the continuity of these interventions and there are evidences proving the opposite, positive changes in clinical outcomes as diabetes, blood pressure and elevated blood cholesterol. In addition some measures as BMI, anthropometric, fitness level have shown good association as prediction of development of chronic disease with low cost (Dishman 2004).

ELIGIBILITY:
Inclusion Criteria The inclusion criteria for participation of these study were never participated of and quality of life and health intervention program at work and had an interest in participating in the study. Included workers ≥ 18years who had to work in the office position, sitting at the computer most of the work shift.

Exclusion criteria: temporary workers and freelancers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Grande, PhD, Principal Investigator — Universidade Metodista de Piracicaba
Locations (1):
- Universidade Metodista de Piracicaba, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data are available when required

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Administrative workplace
Groups:
- Exercise in the Workplace and Educational Intervention: Company A received exercise in the workplace, posters with tips on health and quality of life computer software
  Exercise, Educational Intervention: Exercise were prescribed three times a week with duration of fifteen minutes for three months.
  Educational Intervention were composed by a quality of life computer software and poster with tips on health behaviors
- Exercise in the Workplace: Exercise in the workplace was prescribed three times per week with fifteen minutes of duration. The exercises were mild.
  Exercise, Educational Intervention: Exercise were prescribed three times a week with duration of fifteen minutes for three months.
  Educational Intervention were composed by a quality of life computer software and poster with tips on health behaviors
- Educational Intervention: This company received a quality of life software and poster with tips on health lifestyle.
  Exercise, Educational Intervention: Exercise were prescribed three times a week with duration of fifteen minutes for three months.
  Educational Intervention were composed by a quality of life computer software and poster with tips on health behaviors
- Control Company: No intervention. Control group received no intervention during study period
Period: Overall Study
Arm/Group | Exercise in the Workplace and Educational Intervention | Exercise in the Workplace | Educational Intervention | Control Company
Started | 65 | 62 | 39 | 24
Completed | 60 | 54 | 38 | 20
Not Completed | 5 | 8 | 1 | 4
Not completed — Lost to Follow-up | 5 | 8 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Exercise in the Workplace and Educational Intervention: Participants received exercise in the workplace and educational intervention
- Exercise in the Workplace: Participants received exercise only
- Educational Intervention: Participants received educational intervention only
- Control Company: Participants did not receive any intervention
- Total: Total of all reporting groups
Arm/Group | Exercise in the Workplace and Educational Intervention | Exercise in the Workplace | Educational Intervention | Control Company | Total
Number analyzed (Participants) | 65 | 62 | 39 | 24 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 65 | 62 | 39 | 24 | 190
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (3.54) | 23.9 (5.23) | 28.6 (7.57) | 27.2 (7.7) | 26 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 33 | 15 | 5 | 97
  Male | 21 | 29 | 24 | 19 | 93
Region of Enrollment [Number; unit: participants]
  Brazil | 65 | 62 | 39 | 24 | 190

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life
Description: The instrument contains 80 questions, of which 67 were structured in 5 points Lickert Scale. QVS-80 has four domains: Health Domain (Health) Physical activity (PA), occupational environment domain (AO) and perception of QoL (QOL). The health domain is composed of 30 questions, and the thirteen initial questions refer to history of the existence of chronic diseases such as hypertension, diabetes, obesity, dyslipidemias, bronchitis, allergic rhinitis and cancer; the remaining questions relate to lifestyle and living habits, such as quality of sleep, smoking and consumption of alcohol. The domain of physical activity consists of 15 questions on physical activity. The Domain workplace consists of 11 questions about the physical activity at work and occupational environment. The Domain perception of QoL consists of 24 questions about personal characteristics, and autonomy. The syntax of QVS-80 put the results in a scale of 0 -100 points (the higher the better).
Time Frame: The participants were followed for 3 months
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Exercise in the Workplace and Educational Intervention | Exercise in the Workplace | Educational Intervention | Control Company
Number analyzed (Participants) | 60 | 54 | 38 | 20
units on a scale | 71.5 (3.1) | 68.5 (3.0) | 72 (4.0) | 72 (3.3)

2. Secondary Outcome: Physical Activity Level
Description: The level of physical activity was evaluated by the questionnaire of quality of life. (QVS-80). The physical activity domain is composed of 15 questions considering the ammount of physical activity practiced during leisure time. The instrument is structured in 5 points Lickert Scale. The syntax of QVS-80 put the results in a scale of 0 -100 points (the higher the better).
Time Frame: The participants were followed for 3 months
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Exercise in the Workplace and Educational Intervention | Exercise in the Workplace | Educational Intervention | Control Company
Number analyzed (Participants) | 60 | 54 | 38 | 20
units on a scale | 30 (3.5) | 27 (3.1) | 36 (7.2) | 36 (8.2)

3. Secondary Outcome: Occupational Environment
Description: The occupational environment was assessed by the quality of life questionnaire. (QVS-80). It considers physical aspects like accessibility and psycologic aspects such as stress. The domain consists of 11 questions about occupational environment. The syntax of QVS-80 put the results in a scale of 0 -100 points (the higher the better).
Time Frame: The participants were followed for 3 months
Measure: Median (Standard Deviation); unit: units on a scale 0-100
Arm/Group | Exercise in the Workplace and Educational Intervention | Exercise in the Workplace | Educational Intervention | Control Company
Number analyzed (Participants) | 60 | 54 | 38 | 20
units on a scale 0-100 | 70 (5.3) | 65 (4.2) | 45 (6.5) | 52 (4.2)

4. Secondary Outcome: Changes in Disease Prevalence
Description: the changes in disease prevalence was measured in the same instrument QVS-80. The chronic disease was self-related by the participants.
Time Frame: The participants were followed for 3 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Exercise in the Workplace and Educational Intervention | Exercise in the Workplace | Educational Intervention | Control Company
Number analyzed (Participants) | 60 | 54 | 38 | 20
participants
  Hypertension | 2 [0 to 2] | 2 [0 to 2] | 1 [0 to 1] | 5 [0 to 5]
  Overweight | 11 [0 to 11] | 14 [0 to 14] | 16 [0 to 16] | 8 [0 to 8]
  Dislipedemy | 3 [0 to 3] | 6 [0 to 6] | 1 [0 to 1] | 0 [0 to 0]
  Asthma | 2 [0 to 2] | 11 [0 to 11] | 6 [0 to 6] | 3 [0 to 3]
  Thyreopathy | 2 [0 to 2] | 3 [0 to 3] | 2 [0 to 2] | 0 [0 to 0]

5. Secondary Outcome: Pain Perception
Description: Pain perception were evaluated by the diagram of pain proposed by Corlett in 1995. The part of body which had pain were indicated by the participant. The data were analysed as "yes" or "no" and reported as Odds ratio.
Time Frame: The participants were followed for 3 months
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Exercise in the Workplace and Educational Intervention | Exercise in the Workplace | Educational Intervention | Control Company
Number analyzed (Participants) | 60 | 54 | 38 | 20
Odds Ratio | 2.29 [0.87 to 5.99] | 3.74 [1.16 to 12.02] | 0.94 [0.38 to 2.34] | 1.07 [0.34 to 3.27]

ADVERSE EVENTS:
Time Frame: data were collected after 3 months.
Description: Number of Events Definition: Number of occurrences, in each arm/group, of the adverse event being reported
  None adverse events were reported by any worker in this research
Arm/Group | Exercise in the Workplace and Educational Intervention | Exercise in the Workplace | Educational Intervention | Control Company
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/62 | 0/39 | 0/24
Other Adverse Events (participants affected / at risk) | 0/65 | 0/62 | 0/39 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No